CLINICAL TRIAL: NCT03526419
Title: Pharmacokinetics and Breast Milk Excretion of Liposomal Bupivacaine After TAP Block in Patients Undergoing Cesarean Section Delivery
Brief Title: Exparel PK and Breast Milk Excretion
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003258
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Milk Expression, Breast
Keywords: Liposomal bupivacaine; TAP block; cesarean section
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Bupivacaine liposome — blood and milk samples will be obtained from those subjects after TAP block

SUMMARY:
Investigate the pharmacokinetics of Liposomal Bupivacaine and its excretion in breast milk in patients undergoing TAP block after their scheduled C -section delivery

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women >18 year old, scheduled for elective Cesarean delivery and who desire to have a TAP block performed after delivery.
2. American Society of Anesthesiologists physical status I, II, and III

Exclusion Criteria:

1. Patient refusal or inability to cooperate.
2. Allergy, hypersensitivity, intolerance, or contraindication to liposomal bupivacaine.
3. Severely impaired renal or hepatic function (eg, serum creatinine level >2 mg/dL [176.8 µmol/L], blood urea nitrogen level >50 mg/dL [17.9 mmol/L], serum aspartate aminotransferase [AST] level >3 times the upper limit of normal [ULN], or serum alanine aminotransferase [ALT] level >3 times the ULN).
4. Participants at an increased risk for bleeding or with any coagulation disorder (defined as platelet count less than 80, 000 × 103/mm3 or international normalized ratio greater than 1.5) (all contraindications to TAP block).
5. Clinically significant medical disease in either the mother or baby that, in the opinion of the investigator, would make participation in a clinical study inappropriate. This includes any psychiatric or other disease in the mother that would constitute a contraindication to participation in the study or cause the mother to be unable to comply with the study requirements.
6. Patient membership in a vulnerable population such as a prisoner, mentally unable to provide direct consent etc.
7. Participant has contraindication to breastfeeding or not planning to breastfeed the first 2-3 days after delivery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients undergoing scheduled C-section delivery
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
milk plasma ratio | 72 hours
  AUC for the milk/plasma drug ratio

SECONDARY OUTCOMES:
AUC of plasma | 72 hours
  AUC for drug concentration in plasma
AUC of milk | 72 hours
  AUC for drug concentration in milk

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mustafa HJ, Wong HL, Al-Kofahi M, Schaefer M, Karanam A, Todd MM. Bupivacaine Pharmacokinetics and Breast Milk Excretion of Liposomal Bupivacaine Administered After Cesarean Birth. Obstet Gynecol. 2020 Jul;136(1):70-76. doi: 10.1097/AOG.0000000000003886. PMID 32541292